CLINICAL TRIAL: NCT03571893
Title: Randomized Controlled Trial of an International Commercial Program on Weight Loss and Health Outcomes
Brief Title: Study of an International Commercial Program on Weight Loss and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1026
Record Dates: First submitted 2018-06-01; First posted 2018-06-28 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Weight Loss; Weight Change, Body; Obesity; Diet Modification
MeSH Terms: conditions — Weight Loss; Body Weight Changes; Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions, with assessments occurring prior to randomization, at 3 months and 12 months. Participants will be referred to either Weight Watchers or provided DIY resources. Study staff will not deliver intervention.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to participant treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Watchers Freestyle (Flex) (Experimental): Participate in Commercially Available behavioral weight loss program delivered by Weight Watchers International in the community
  Interventions: Behavioral: Weight Watchers Freestyle (Flex)
- DIY Personal Plan (Active Comparator): Receive informational resources for healthy lifestyle change to promote weight loss
  Interventions: Behavioral: DIY Personal Plan

INTERVENTIONS:
Behavioral: Weight Watchers Freestyle (Flex) — Participants will be referred to their local Weight Watchers meeting and provided with a promotional code to allow them to participate in the Weight Watchers program free of charge for 12 months. At the randomization visit, study staff will help participants identify a convenient Weight Watchers meeting location and download the program app onto their smartphone.
  Arms: Weight Watchers Freestyle (Flex)
Behavioral: DIY Personal Plan — Participants will be provided with a written resource with descriptions of a variety of approaches that have been shown to promote healthy weight loss through behavioral modification. Participants will be encouraged to assess their preferences for dietary change and physical activity and adopt an approach that will lead to negative energy balance and moderate (1-2 lbs. per week) weight loss.
  Arms: DIY Personal Plan

SUMMARY:
This study is a randomized controlled trial (RCT) of the Weight Watchers (WW) Freestyle ® (Flex® in UK) weight loss program compared to a control group following a do-it-yourself (DIY) approach for 12 months. Participants in the United States, Canada and the UK (n=360 total) will be randomly assigned to either participate in the commercially available WW program in their local community or to follow their own approach for weight loss. This study will examine the impact of the WW program on weight, fitness levels, quality of life, health behaviors and other health outcomes in overweight and obese adults after 3 and 12 months.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of the Weight Watchers program delivered in the community to a DIY approach for weight loss.

Potential participants will be recruited through a variety of advertisement methods. Those individuals responding to these advertisements will undergo web-based preliminary screening. Initially eligible individuals will be contacted by phone to receive more detailed information and to complete screening. Eligible and interested participants will be consented in person and complete screening assessments that will be used to confirm eligibility (height and weight to determine body mass index, resting blood pressure. For participants deemed to be eligible and randomized to participate in this study, these measures will also be used as their baseline data from analysis. Additional data collection will be collected at the baseline assessment visit, with assessments repeated at 3 months and after the intervention at 12 months. Assessments will include the following:

Height and Weight Resting Blood Pressure and Heart Rate Aerobic Stamina Flexibility Waist Circumference Dietary Intake Additional Questionnaires to assess demographics, sleep, food cravings, hunger and satiety, weight control strategies, affect, lifestyle activities

Group assignment will be revealed to study participants in a separate visit/contact after all assessment procedures and randomization is completed. The contact will last 15-30 minutes and participants will be provided with the resources they need to either follow the Weight Watchers program or the DIY approach. The Weight Watchers orientation and DIY intervention will not be provided by staff who collect measurements in order to preserve the blinding of the measurement staff. Following randomization reveal, the staff will maintain communication in order to promote retention (e.g., birthday card or small token reinforcer such as a water bottle sent to all participants).

WEIGHT WATCHERS FREESTYLE (FLEX) GROUP Intervention Description Participants randomized to the WW Freestyle (Flex) treatment arm will be referred to their local WW Meetings + Online Plus program delivered at a WW center / meeting convenient to them. At the randomization visit, they will be provided with a code to sign up for the Weight Watchers program free of charge for 12 months. They will also be guided to download the smartphone app on their phone, provided with a list of local meetings, and instructed on how to start the Weight Watchers intervention.

The following describes the weight loss intervention that is delivered solely through the commercially available Weight Watchers program. Measurement staff will not be involved in delivery of this intervention.

Program type. Participants will receive a program with a structured, lifestyle modification, weight-loss methodology. Specifically, it will include 1) a food plan, which is based on balanced diet and healthy eating, 2) an activity plan, designed to promote progressive physical activity increase, 3) group support, and 4) cognitive behavior modification. Participants will determine their weight goal and will be encouraged to utilize all intervention components.

Beyond the Scale. This holistic and personalized program focuses on multiple ways for participants to define success, on and off the scale. The three main components are: eating healthier, moving more, and finding and shifting the study subject's mindset.

Weekly meetings. Weight Watchers members attend weekly Weight Watchers meetings conducted in local commercial centers with a group Leader and a receptionist and last30-60 minutes. Meetings consist of lesson delivery of a new behavioral skill or knowledge transfer on healthy habits, check-ins with each participant on their previous week, and group discussions on the week's topic and application of that skill in their own lives. The discussions are led by Weight Watchers Leaders, who are Lifetime members who have successfully achieved and maintained a healthier body weight through the Weight Watchers program, and have successfully completed a leader skills training course and ongoing professional development and quality assurance (QA). WW participants have their weight measured at each meeting on regularly calibrated scales.

Intervention materials. Weight Watchers participants receive: 1) access to an app for food and activity tracking, 2) welcome packet a menu of 'how to's' and inspiration to get started and weekly lesson plans delivered by the Meeting Leader, 3) weekly take-home skill builder worksheet and content within the app 4) Weight Watchers emails, and 4) access to social support from other WW Leaders and WW members through on online support portal.

Dietary goals. Dietary plan. The core of the Food Program is the SmartPoints® weight loss system, which is a method of self-monitoring dietary intake. The SmartPoints system assigns each food and beverage a SmartPoints value per portion based on its nutrition, factoring in four components: calories, sugar, saturated fat, and protein. SmartPoints encourages a healthier pattern of eating. This is translated into the following general guidelines: certain foods have a SmartPoints value of zero which includes plant-based proteins, skinless chicken and turkey breast, eggs, non-fat yogurt, skinless fish, fruits and most vegetables (excludes starchy vegetables). For foods outside these categories, foods higher in lean protein, such as lean cuts of steak and ham, have lower SmartPoints values while foods higher in unhealthy saturated fats and sugar have higher Smartpoints values

SmartPoints Budget. Based on the Mifflin St-Jeor formula, which factors in age, gender, height, and weight, participants will get a personalized SmartPoints Budget. The SmartPoints budget consists of: a daily SmartPoints Target plus an extra bank of Weekly SmartPoints for flexibility. Participants are free to spend their SmartPoints however they wish and can 'roll over' up to 4 SmartPoints a day into their weeklies for added flexibility.

Food Log. Participants will be encouraged to track their SmartPoints each day on the Weight Watchers app provided to them. Within the app there is a wealth of tools to help find and track food choices, which includes; a barcode scanner to quickly identify foods, recipes, restaurant and grocery store items in a database.

Activity goals. FitPoints. A large part of the Beyond the Scale program is the FitPoints™ system, which is a method of self-monitoring physical activity. The FitPoints system assigns each activity a FitPoint value based on its duration (minutes) and intensity based on a participant's current weight and FitPoints emphasizes activity because it feels good, not solely as a means to swap for SmartPoints. FitPoints highlights that all activity counts and adds up; "some is better than none".

FitPoints goal. Participants will receive a personalized daily FitPoints goal based on their fitness level and goals.

Activity Log Participants will be encouraged to track their FitPoints each day on the Weight Watchers app provided to them.

Mindset Approach. The Weight Watchers Freestyle/Flex program promotes the adoption of skills and techniques to adopt a positive mindset in order to support lifestyle change and healthy weight Participants receive digital and print materials around these topics and in person support in the meetings.

DO-IT-YOURSELF GROUP Participants randomized to the DIY group will be provided with a brief resource guide with basic information about a variety of healthful behavioral weight loss approaches (meal plans, apps for calorie tracking, meal replacements, dietary approaches to reduce calories healthfully such as following a low fat or low carb diet, and moderate physical activity) and encouraged to choose an approach that would fit with their lifestyle. The resource guide will provide model "profiles" of lifestyle factors that may help the individual choose the approach that would work best for them. These approaches are consistent with information that can be found in the general press and will be limited to approaches that are deemed healthful by weight loss and medical professionals. Participants will be informed that many people follow a DIY approach and can be successful (will reference the National Weight Control Registry which is a research-based registry of individuals who have lost weight and kept is off successfully; 50% of whom followed a DIY approach). For retention, participants in the DIY group will be notified that if they choose to utilize WW after the completion of the study, they will be offered free vouchers for 12 months of the WW program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18-75 years
* With or without previous WW experience
* Self-reported height/weight resulting in a Body Mass Index (BMI) of 25 to 45 (will be confirmed at the Baseline Assessment visit).
* Self report that he/she feels the need to lose weight.
* Willing to discontinue any current over-the-counter (OTC) supplements not recommended/prescribed by physician, with the exception of multivitamins or other vitamin supplement.
* Willing to be randomized to one of two groups and follow recommendations according to study protocol.
* Willing to include demographic information (e.g., ethnicity, income and education).
* Use of a personal smartphone (iOS 9.0 or Android 4.1)
* The willingness and ability to download, navigate and use applications on their smartphone on a daily basis (minimum training will be provided)
* Ability to commit to attending study assessment visits at 0, 3 and 12 months
* Residing within 30 miles of a study assessment location
* Read, write and speak English

Exclusion Criteria:

* Participants that were a member of Weight Watchers within the past 12 months.
* Unwilling to refrain from using Weight Watchers if assigned to the DIY group.
* Participants that are involved in any other research studies at this time (also, cannot join other research studies while in this study, over the next 12 months) that would interfere with their ability to adhere to the protocol (i.e., attend assessment visits, attend WW meetings).
* Given birth past six months, currently pregnant, or planning on becoming pregnant over the next 12 months.
* Weight loss of ≥ 5 kg in the previous 6 months (and kept > 5 kg off).
* Ever been diagnosed with an eating disorder (anorexia nervosa, bulimia).
* Reported health problems that make weight loss or unsupervised exercise unsafe or unreasonable (e.g., orthopedic limitations, heart problems)
* Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months.
* Taking any prescription medication with known effects on appetite or weight (e.g., oral steroids, weight loss medications such as Qsymia, Contrave, etc.) with the exception of subjects on a stable dose of Selective serotonin reuptake inhibitors (SSRIs) for 6 months
* Currently have chronic/inflammatory gastrointestinal disorder (irritable bowel syndrome acceptable).
* History of heart problems (e.g., angina, bypass surgery, myocardial infarction, etc.) within previous 6 months.
* Resting systolic blood pressure >160 mmHg or resting diastolic blood pressure >100 mmHg (confirmed at baseline visit)
* Currently have type 1 or type 2 diabetes
* Ever had surgical procedure for weight loss.
* Major surgery within the previous 6 months that would interfere with consuming a regular diet and performing physical activity such as walking.
* Presence of implanted cardiac defibrillator or pacemaker.
* History of cancer within past 5 years or current treatment for cancer (completely resected basal or squamous cell carcinoma acceptable if treatment completed more than 6 months prior to enrollment).
* Hospitalization for psychiatric problems during the past 12 months
* Planning to relocate in the next 12 months
* Another member of the household is participating in this research study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Change in Weight from Baseline to Month 12 | Baseline, Month 12
  Weight will be measured in kg on a digital scale

SECONDARY OUTCOMES:
Change in weight from Baseline to Month 3 | Baseline, Month 3
  Weight will be measured in kg on a digital scale
Change in Body Mass Index (BMI) from Baseline to Month 3 | Baseline, Month 3
  BMI in kg/m²
Change in Body Mass Index (BMI) from Baseline to Month 12 | Baseline, Month 12
  BMI in kg/m²
Percent weight change at Month 3 | Month 3
  Percent of baseline weight lost or gained
Percent weight change at Month 12 | Month 12
  Percent of baseline weight lost or gained
Change in Blood pressure from Baseline to Month 3 | Baseline, Month 3
  Systolic and diastolic blood pressure will be measured in mmHg after a 5 minute rest
Change in Blood pressure from Baseline to Month 12 | Baseline, Month 12
  Systolic and diastolic blood pressure will be measured in mmHg after a 5 minute rest
Change in resting pulse from Baseline to Month 3 | Baseline, Month 3
  Pulse will be measured in beats per minute after a 5 minute rest
Change in resting pulse from Baseline to Month 12 | Baseline, Month 12
  Pulse will be measured in beats per minute after a 5 minute rest
Change in Sleep Scores from Baseline to Month 3 | Baseline, Month 3
  Pittsburgh Sleep Quality Index (PSQI): Measures sleep disturbance and usual sleep habits during the prior month only using seven clinically derived domains of sleep difficulties: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. Global PSQI is a summary of the seven domains. Each Domain is scored from 0 to 3, therefore PSQI has a range of 0 (better) to 21 (worse). Interpretation of the PSQI is that a score less than 5 is associated with good sleep quality and a score of 5 or greater is associated with poor sleep quality.
Change in Sleep Scores from Baseline to Month 12 | Baseline, Month 12
  Pittsburgh Sleep Quality Index (PSQI): Measures sleep disturbance and usual sleep habits during the prior month only using seven clinically derived domains of sleep difficulties: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. Global PSQI is a summary of the seven domains. Each Domain is scored from 0 to 3, therefore PSQI has a range of 0 (better) to 21 (worse). Interpretation of the PSQI is that a score less than 5 is associated with good sleep quality and a score of 5 or greater is associated with poor sleep quality.
Change in Food craving Scores from Baseline to Month 3 | Baseline, Month 3
  The Food Craving Inventory-II (FCI-II) is a validated self-report measure for general cravings and cravings for specific types of foods and will be completed at baseline, Months 3 and 12. Respondents rate the frequency of cravings since the last time they completed the survey for each of 33 food items using a five-point Likert scale (1, never; 2, rarely; 3, sometimes; 4, often; 5, always/almost every day). The FCI-II consists of 5 scales (sweets, high fats, carbohydrates/starches, fast food fats, and fruits & vegetables) that constitute the higher order construct of food cravings (the total score).
Change in Food craving Scores from Baseline to Month 12 | Baseline, Month 12
  The Food Craving Inventory-II (FCI-II) is a validated self-report measure for general cravings and cravings for specific types of foods and will be completed at baseline, Months 3 and 12. Respondents rate the frequency of cravings since the last time they completed the survey for each of 33 food items using a five-point Likert scale (1, never; 2, rarely; 3, sometimes; 4, often; 5, always/almost every day). The FCI-II consists of 5 scales (sweets, high fats, carbohydrates/starches, fast food fats, and fruits & vegetables) that constitute the higher order construct of food cravings (the total score).
Change in VAS Scores for Hunger and fullness from Baseline to Month 3 | Baseline, Month 3
  The most commonly used tool to measure subjective sensations of hunger is the Visual Analogue Scale (VAS). A VAS measures sensations that range across a continuum of values and cannot be easily directly measured. Operationally, the VAS is a horizontal line measuring exactly 100 mm in length, anchored by word descriptors (i.e., 0=Not at all hungry, 100=Extremely hungry) at each end. At baseline, Months 3 and 12, participants will be asked to complete a three item VAS by placing a mark on the line at the point they feel represents their response to the question.
Change in VAS Scores for Hunger and fullness from Baseline to Month 12 | Baseline, Month 12
  The most commonly used tool to measure subjective sensations of hunger is the Visual Analogue Scale (VAS). A VAS measures sensations that range across a continuum of values and cannot be easily directly measured. Operationally, the VAS is a horizontal line measuring exactly 100 mm in length, anchored by word descriptors (i.e., )0=Not at all hungry, 100=Extremely hungry) at each end. At baseline, Months 3 and 12, participants will be asked to complete a three item VAS by placing a mark on the line at the point they feel represents their response to the question.
Change in weight control strategies used from Baseline to Month 3 | Baseline, Month 3
  The Weight Control Strategies Scale (WCSS) is a 30 item self-report measure of behavioral strategies commonly used for weight loss and will be used to measure strategies used for the purpose of weight loss. The measure was validated in a pooled sample from three behavioral weight loss trials. Principal components analysis with varimax rotation revealed a four-component solution for the WCSS, representing the following subscales: Dietary Choices, Self-monitoring Strategies, Physical Activity, and Psychological Coping (α from 0.79 to 0.89). Longitudinal analyses showed that WCSS subscale scores increased during treatment (P < 0.01). In adjusted models, changes in WCSS total and subscale scores were associated with post-treatment weight loss (P < 0.01). Higher scores indicate more strategies endorsed and subscales indicate the type of strategies. Higher scores are predictive of weight loss.
Change in weight control strategies used from Baseline to Month 12 | 12 months
  The Weight Control Strategies Scale (WCSS) is a 30 item self-report measure of behavioral strategies commonly used for weight loss and will be used to measure strategies used for the purpose of weight loss. The measure was validated in a pooled sample from three behavioral weight loss trials. Principal components analysis with varimax rotation revealed a four-component solution for the WCSS, representing the following subscales: Dietary Choices, Self-monitoring Strategies, Physical Activity, and Psychological Coping (α from 0.79 to 0.89). Longitudinal analyses showed that WCSS subscale scores increased during treatment (P < 0.01). Higher scores indicate more strategies endorsed and subscales indicate the type of strategies. Higher scores are predictive of weight loss.
Change in Dietary intake Score from Baseline to Month 3 | Baseline, Month 3
  Diet intake will be measured using the Yale 24hr Food Frequency Questionnaire (FFQ), which is a brief nutrition self-monitoring tool measuring the intakes of fruits and vegetables, percentage energy from fat, and fiber, by focusing on specific foods consistently linked to weight gain or loss. Participants are asked to recall food consumption of various categories over 24-hour periods. The survey is currently being validated.
Change in Happiness Scores from Baseline to Month 3 | 3 months
  Participants will be asked to complete the Oxford Happiness Questionnaire (OHQ)at baseline, Months 3 and 12. The OHQ is a validated self-report measure for broad personal happiness. Respondents rate 29 sentences on a 6 point Likert scale (1, strongly disagree; 6, strong agree).
Change in Dietary intake Score from Baseline to Month 12 | Baseline, Month 12
  Diet intake will be measured using the Yale 24hr FFQ, which is a brief nutrition self-monitoring tool measuring the intakes of fruits and vegetables, percentage energy from fat, and fiber, by focusing on specific foods consistently linked to weight gain or loss. Participants are asked to recall food consumption of various categories over 24-hour periods. The survey is currently being validated.
Change in Happiness Scores from Baseline to Month 12 | Baseline, Month 12
  Participants will be asked to complete the Oxford Happiness Questionnaire (OHQ) at baseline, Months 3 and 12. The OHQ is a validated self-report measure for broad personal happiness. Respondents rate 29 sentences on a 6 point Likert scale (1, strongly disagree; 6, strong agree).
Change in Quality of Life Score from Baseline to Month 3 | Baseline, Month 3
  The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a validated self-report measure for an individual's perception of how their weight affects their day-to-day life and will be completed at baseline, Months 3 and 6. Respondents rate the degree to which their weight affects them on 31 items using a five-point Likert scale (1, never true; 2, rarely true; 3, sometimes true; 4, usually true; 5, always true). The IWQOL-Lite consists of 5 scales (physical function, self-esteem, sexual life, public distress, and work).
Change in Quality of Life Score from Baseline to Month 12 | Baseline, Month 12
  The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a validated self-report measure for an individual's perception of how their weight affects their day-to-day life and will be completed at baseline, Months 3 and 6. Respondents rate the degree to which their weight affects them on 31 items using a five-point Likert scale (1, never true; 2, rarely true; 3, sometimes true; 4, usually true; 5, always true). The IWQOL-Lite consists of 5 scales (physical function, self-esteem, sexual life, public distress, and work).
Change in Positive and Negative affect Score from Baseline to Month 3 | 3 months
  The Scale of Positive and Negative Experience (SPANE) is a brief 12-item scale, with six items corresponding to positive emotions and six items corresponding to negative emotions. Each item is scored on a scale ranging from 1 to 5, where 1 represents "very rarely or never" and 5 represents "very often or always." The positive and negative scales are scored separately and each range from 6 to 30. The two scores can also be combined as a scale of balanced affect. Internal consistency is good (ranging from 0.81-0.89 across the scales), as is temporal stability (0.62-0.68). The SPANE has performed well in terms of convergent validity with other measures of emotion, well-being, happiness, and life satisfaction.
Change in Positive and Negative affect Score from Baseline to Month 12 | Baseline, Month 12
  The SPANE is a brief 12-item scale, with six items corresponding to positive emotions and six items corresponding to negative emotions. Each item is scored on a scale ranging from 1 to 5, where 1 represents "very rarely or never" and 5 represents "very often or always." The positive and negative scales are scored separately and each range from 6 to 30. The two scores can also be combined as a scale of balanced affect. Internal consistency is good (ranging from 0.81-0.89 across the scales), as is temporal stability (0.62-0.68). The SPANE has performed well in terms of convergent validity with other measures of emotion, well-being, happiness, and life satisfaction.
Change in Health-Promoting Lifestyle Practices Score from Baseline to Month 3 | 3 months
  The Health Promoting Lifestyle Profile II (HPLP-II) is a 52-item instrument measuring self-initiated health behaviors that serve to maintain or enhance the level of self-actualization and wellness. Included are six subscales: physical activity, spiritual growth, health responsibility, interpersonal relations, nutrition, and stress management. It is self-administered and uses a 4-point response format yielding a score for overall health-promoting lifestyle which is obtained by calculating a mean of the individual's responses to all 52 items. Similarly, subscale scores are obtained by calculating a mean of the responses to subscale items. Scores range from 1 = Never to 4 = Routinely, with a higher score corresponding to a more health-promoting lifestyle.
Change in Health-Promoting Lifestyle Practices Score from Baseline to Month 12 | Baseline, Month 12
  The Health Promoting Lifestyle Profile II (HPLP-II) is a 52-item instrument measuring self-initiated health behaviors that serve to maintain or enhance the level of self-actualization and wellness. Included are six subscales: physical activity, spiritual growth, health responsibility, interpersonal relations, nutrition, and stress management. It is self-administered and uses a 4-point response format yielding a score for overall health-promoting lifestyle which is obtained by calculating a mean of the individual's responses to all 52 items. Similarly, subscale scores are obtained by calculating a mean of the responses to subscale items. Scores range from 1 = Never to 4 = Routinely, with a higher score corresponding to a more health-promoting lifestyle.
Change in Flexibility from Baseline to Month 3 | Baseline, Month 3
  Flexibility will be measured using the sit-and-reach test. They will then sit on the floor with their legs outstretched in front of them and their feet perpendicular to the floor (toes facing up). A vertical 12 inch box will be placed against their feet. The participant will then be asked to place one hand over the other such that the tops of their two middle fingers will be on top of one another. Finally, the participant will be instructed to slowly stretch forward and slide their fingers along the box as far as possible. A ruler is used to measure the distance they can reach. This test is repeated three times and the best score will be retained.
Change in Flexibility from Baseline to Month 12 | Baseline, Month 12
  Flexibility will be measured using the sit-and-reach test. They will then sit on the floor with their legs outstretched in front of them and their feet perpendicular to the floor (toes facing up). A vertical 12 inch box will be placed against their feet. The participant will then be asked to place one hand over the other such that the tops of their two middle fingers will be on top of one another. Finally, the participant will be instructed to slowly stretch forward and slide their fingers along the box as far as possible. A ruler is used to measure the distance they can reach. This test is repeated three times and the best score will be retained.
Change in Aerobic stamina from Baseline to Month 3 (walk test) | 3 months
  Aerobic stamina will be measured using the six minute walk test and the one-minute sit to stand test. Aerobic Capacity: Participants will complete a 6 minute walk test on a designated walking course. The 6 minute walk test is a measure of functional and aerobic capacity. Participants are asked to walk at a brisk, yet comfortable pace for a total of 6 minutes. Distance covered in 6 minutes, pre and post perceived exertion and breathlessness and post test pulse are measured.
Change in Aerobic stamina from Baseline to Month 12 (walk test) | Baseline, Month 12
  Aerobic stamina will be measured using the six minute walk test and the one-minute sit to stand test. Aerobic Capacity: Participants will complete a 6 minute walk test on a designated walking course. The 6 minute walk test is a measure of functional and aerobic capacity. Participants are asked to walk at a brisk, yet comfortable pace for a total of 6 minutes. Distance covered in 6 minutes, pre and post perceived exertion and breathlessness and post test pulse are measured.
Change in exercise capacity from baseline to 3 months (sit to stand test) | Baseline, Month 3
  Exercise capacity will be measured using the one-minute sit to stand test. The test measures the number of times a participant can rise from a seated position with arms crossed over chest during a one minute period.
Change in exercise capacity from Baseline to 12 months (sit to stand test) | Baseline, Month 12
  Exercise capacity will be measured using the one-minute sit to stand test. The test measures the number of times a participant can rise from a seated position with arms crossed over chest during a one minute period.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F. Tate, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States
- Canada (2):
  - University of British Columbia-Okanagan, Kelowna, British Columbia
  - University of British Columbia-Vancouver, Vancouver, British Columbia
- University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tate DF, Lutes LD, Bryant M, Truesdale KP, Hatley KE, Griffiths Z, Tang TS, Padgett LD, Pinto AM, Stevens J, Foster GD. Efficacy of a Commercial Weight Management Program Compared With a Do-It-Yourself Approach: A Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2226561. doi: 10.1001/jamanetworkopen.2022.26561. PMID 35972742